CLINICAL TRIAL: NCT05172908
Title: The Effect of Preoperative Intravenous Dexamethasone on Postoperative Rebound Pain and Sleep Quality in Patients Receiving Ultrasonography-Guided Ilioinguinal and Iliohypogastric Nerve Block for Inguinal Hernia Repair
Brief Title: The Effect of Dexamethasone on Rebound Pain in Patients Receiving Ilioinguinal and Iliohypogastric Nerve Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karaman Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08-2021/11
Record Dates: First submitted 2021-12-10; First posted 2021-12-29 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2022-12

CONDITIONS: Inguinal Hernia
Keywords: Dexamethasone; Ilioinguinal and Iliohypogastric nerve block; Bupivacaine; Rebound Pain
MeSH Terms: conditions — Hernia, Inguinal | interventions — Dexamethasone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Dexa (Active Comparator): After induction of general anesthesia, an ultrasound-guided block of the ilioinguinal and iliohypogastric nerve block will be performed using 20 ml 0.5% bupivacaine. 5 mg dexamethasone in a 50 ml syringe containing normal saline will be infused within 15 minutes. A multimodal analgesia regimen will be applied postoperatively.
  The syringe will be prepared by a nurse outside the research team and the study participants, care providers, and data collectors will be blinded to the allocation throughout the study
  Interventions: Drug: Dexamethasone
- Group S (Sham Comparator): After induction of general anesthesia, an ultrasound-guided block of the ilioinguinal and iliohypogastric nerve block will be performed using 20 ml 0.5% bupivacaine. 50 mL normal saline in a 50 ml syringe will be infused within 15 minutes. A multimodal analgesia regimen will be applied postoperatively.
  The syringe will be prepared by a nurse outside the research team and the study participants, care providers, and data collectors will be blinded to the allocation throughout the study
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Dexamethasone — 5 mg dexamethasone in a 50 ml syringe containing normal saline will be infused within 15 minutes.
  The syringe will be prepared by a nurse outside the research team and the Study participants, care providers, and data collectors will be blinded to the allocation throughout the study.
  Global Quality of Recovery- 15 score and standard pain follow-up scores will be noted.
  Other Names: Global Quality of Recovery-15 score; Standard Pain Follow up
  Arms: Group Dexa
Drug: Saline — A 50 ml syringe containing normal saline will be infused within 15 minutes. The syringe will be prepared by a nurse outside the research team and the study participants, care providers, and data collectors will be blinded to the allocation throughout the study.
  Global Quality of Recovery- 15 score and standard pain follow-up scores will be noted.
  Other Names: Global Quality of Recovery-15 score; Standard Pain Follow up and Monitorization
  Arms: Group S

SUMMARY:
Rebound pain is a newly defined phenomenon, observed within the first 24 hours after the operation. Open inguinal hernia repair is a common surgical procedure that can be associated with pain of the either acute or chronic character. A peripheral nerve block of the ilioinguinal (IIN) and iliohypogastric (IHN) nerves is a relatively well-known method for postoperative pain management. However, rebound pain after IIN/IHN block resolution may reduce its overall benefit. The primary aim is to assess whether intravenous dexamethasone reduces postoperative opioid consumption and the incidence of rebound pain in patients undergoing unilateral hernia repair in adults.

DETAILED DESCRIPTION:
Male patients older than 18 years, of American Society of Anesthesiologists physical status I or II, and scheduled for unilateral primary hernia repair with a Lichtenstein style (open surgery with insertion of mesh) under general anesthesia will be included in the study. The patients will be randomized using a computer-generated randomization technique. After induction of general anesthesia, the patients in the dexamethasone group (Group Dex) will receive 5 mg dexamethasone in a 50 ml syringe containing normal saline. The patients in the saline group (Group S) will receive normal saline in a 50 ml syringe. Ultrasound-guided block of the ilioinguinal (IIN) and iliohypogastric (IHN) nerves will be performed on all patients included in both groups. The primary aim is to assess whether intravenous dexamethasone reduces postoperative opioid consumption and the incidence of rebound pain in patients undergoing unilateral hernia repair in adults.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* Having signed a written informed consent form
* Scheduled for unilateral primary hernia repair Lichtenstein style (open surgery with insertion of mesh) under general anesthesia

Exclusion Criteria:

* Chronic opioid use (more than one month of 60 mg of oral morphine equivalents daily)
* Contraindications to peripheral nerve blocks including localized infection, coagulopathy, or allergy to local anesthetics
* Stomach ulcer
* Severe obesity (body mass index > 35 kg/m2)
* Uncontrolled Diabetes
* Psychiatric disorders
* Systemic steroid use
* Neuropathic disorder
* Can not communicate in Turkish

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Modified Rebound Pain Score | Postoperative 24 hours
  Modified Rebound Pain score is described as the difference between the last recorded postanesthesia care pain score while it will be working and the highest pain score reported within the first 24 h after IIN/IHN blocks will be performed.
  Pain score will be calculated with Numeric Rating Scale (NRS)(0 = no pain; 10 = worst pain imaginable)
Analgesic consumption | Postoperative 24 hours
  Postoperative total opioid consumption

SECONDARY OUTCOMES:
Numerical Rating Scale scores at rest and mobilization | Postoperative 48 hours
  Pain scores (0 = no pain; 10 = worst pain imaginable) using a Numerical Rating Scale (NRS) ranging from 0 to 10.
Quality of Recovery 15 Score | Postoperative Day 1
  Quality of Recovery (QoR)-15 survey.Minimum value: 0, Maximum value: 150, higher scores mean better.
Quality of Sleep | One week after surgery
  Patient's perceived sleep quality will be assessed with Likert scale.Likert scale is scored from 1(very dissatisfied) to 5 (very satisfied).
Analgesic consumption | Postoperative 48 hours
  Postoperative total opioid consumption
Adverse events | Postoperative 24 hour
  Incidence of nausea and vomiting during postoperative 24 hour time period will be noted.
Glucose measurement | Postoperative 24th hour
  Glucose measurement
Surgical infection | Postoperative 14 days
  Surgical infection

CONTACTS AND LOCATIONS:
Overall Officials: Muhammet Korkusuz, MD, Principal Investigator — Karaman Training and Research Hospital
Locations (1):
- Karaman Taining and Research Hospital, Karaman, Turkey (Türkiye)

REFERENCES:
- [Derived] Korkusuz M, Basaran B, Et T, Bilge A, Yarimoglu R, Kurucay Y. The effects of dexamethasone added to ilioinguinal/iliohypogastric nerve (IIN/IHN) block on rebound pain in inguinal hernia surgery: a randomized controlled trial. Hernia. 2023 Dec;27(6):1571-1580. doi: 10.1007/s10029-023-02841-9. Epub 2023 Jul 21. PMID 37477788